CLINICAL TRIAL: NCT01236690
Title: The Clinical Research of the Intermediate and Advanced Hepatoma Treated by Cinobufacin by Perfusion of Hepatic Artery Combining the Arterial Embolotherapy
Brief Title: Study of Hepatoma Treated by Perfusing Cinobufacin Through Hepatic Artery Combining Embolotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Changquan Ling, Department of TCM, Shanghai Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLing
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-10

CONDITIONS: Hepatoma; Cinobufacin Injection
Keywords: Transcatheter arterial embolization; Cinobufacin injection; hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — huachansu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cinobufacin injection — Cinobufacin by Perfusion of Hepatic Artery Combining the Arterial Embolotherapy
  Other Names: Z34020273

SUMMARY:
Cinobufacini has the effects of anticancer, improving the liver function, elevation of immunity and little side effects, and is important and significant for the patients with hepatitis, liver cirrhosis and hepatomas.

Compared with transarterial chemoembolization (TACE) , the clinical effect of cinobufacini is non-inferior/ equivalent.Compared with TACE, cinobufacini is superior in security .

DETAILED DESCRIPTION:
Inclusion criterion :

1. The sex does not limit, age:18-70 years old .
2. The patients have inoperable advanced hepatoma without serious disorder in liver and renal, tumor occupation< 70 %
3. The patients have failure in surgical intervention or resection operation recidivist
4. Hepatic function Child-pugh A、B
5. All the cases have the definite final diagnosis of imageology results such as MRI、CT 、B ultrasonic or cytology results
6. The patient's prediction of live time>6 months, who can tolerant of TACE and has quality of life ECOG score<3
7. The patients participate the clinical trial voluntarily and have already signed informed consent

Exclusion criterion :

1. Main portal vein was obstructed completely.
2. The occupation of tumor are 70 % or more than 70 % in the whole liver
3. The patient has TACE or other antineoplaston
4. After carcinosectomy the patient has the prophylactic
5. The patient is with renal inadequacy: Cr≥133 umol/L
6. Severe cardiovascular disease
7. The patient is with other diseases to influence the proposal

ELIGIBILITY:
Inclusion Criteria:

1. The sex does not limit, age:18-70 years old ;
2. The patients have inoperable advanced hepatoma without serious disorder in liver and renal, tumor occupation< 70 %;
3. The patients have failure in surgical intervention or resection operation recidivist;
4. Hepatic function Child-pugh A、B;
5. All the cases have the definite final diagnosis of imageology results such as MRI、CT 、B ultrasonic or cytology results ;
6. The patient's prediction of live time>6 months, who can tolerant of TACE and has quality of life ECOG score<3;
7. The patients participate the clinical trial voluntarily and have already signed informed consent.

Exclusion Criteria:

1. Main portal vein was obstructed completely;
2. The occupation of tumour are 70 % or more than 70 % in the whole liver;
3. The patient has recepted TACE or other antineoplaston;
4. After carcinosectomy the patient has the prophylactic;
5. The patient is with renal inadequacy: Cr≥133 umol/L
6. Severe cardiovascular disease;
7. The patient is with other diseases to influence the proposal;
8. All over the body generally have metabasis or be with other malignant neoplastic disease;
9. In the process of participation of other medicinal trial;
10. Gravidity, lactation ,hypersensitiveness constitution or have already known adverse reaction or taboo.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the patient's respondence for the therapy is carried out every phase, according to RECIST:CR,PR,SD and PD. | Nov. 2010 to Nov. 2013
  The evaluation of the patient's respondence for the therapy is carried out every phase, according to RECIST:CR,PR,SD and PD.

CONTACTS AND LOCATIONS:
Overall Officials: Ling chang quan, doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Department of TCM, Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality, China